CLINICAL TRIAL: NCT03429036
Title: Biospecimen Procurement for the Study of Head and Neck Disorders
Brief Title: Biospecimen Procurement for Head and Neck Disorders
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180051; 18-DC-0051
Record Dates: First submitted 2018-02-09; First posted 2018-02-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08-01

CONDITIONS: Hearing Disorder; Oral Mucosal Disease; Pharyngeal Neoplasm; Head and Neck Neoplasms; Laryngeal Disease
Keywords: Genomic DNA; DNA Banking; Tissue Sample; Saliva; Blood Collection; Natural History
MeSH Terms: conditions — Hearing Disorders; Pharyngeal Neoplasms; Head and Neck Neoplasms; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects must be diagnosed with a disorder of the head and neck region

SUMMARY:
Background:

Researchers want to learn more about head and neck disorders. Understanding these disorders could help them find better treatments. To do this, they are collecting tissue samples for research.

Objective:

To create a repository of tissue samples and data to better study conditions of the head and neck.

Eligibility:

People who had or will have tissue samples taken because of a head or neck disorder. They must be ages 3 and older and not pregnant to join Part 2.

Design:

Participants will be screened with a questionnaire, medical history, and physical exam.

Part 1. Participants will give permission for any of their tissue samples leftover from private care or other research protocols to be used.

If participants tissue did not contain normal tissue or if they have a condition that suggests a genetic issue, they will be invited to join Part 2.

Part 2: Participants will have additional samples collected. These could be:

* Blood: Blood is drawn through a needle in the arm.
* Cheek swab or brushing: A cotton swab or small brush is rubbed inside the cheek.
* Saliva: They rinse their mouth with water and spit into a tube or cup.
* Skin biopsy: They are injected with a numbing drug. A biopsy tool removes a small piece of skin.
* Mucosal biopsy: They are injected in the mouth with a numbing medication. A small piece of tissue from the inside of the cheek is removed.

Participants samples will be used for future research, including genetic testing.

DETAILED DESCRIPTION:
Background:

NCI Head and Neck Clinical Research Program (H&N CRP) investigators are studying the natural history and treatment of diverse conditions of the head and neck at the National Institutes of Health (NIH). These studies require the collection of biospecimens for research purposes.

Studies performed may support development of future protocols that include new therapeutic agents, novel treatment approaches, and new prognostic and diagnostic models for individuals with disorders of the head and neck affecting human communication.

Objectives:

-Primary: To create a biorepository of diseased and normal tissue specimens for research purposes from individuals with head and neck disorders.

Eligibility:

* Participants must be diagnosed with a disorder of the head and neck region.
* Age >= 3 years

Design:

* Up to 1000 participants will be enrolled.

  * Part 1: Participants with head and neck disorders will be asked to share waste material from surgical procedures to create a biorepository of diseased and normal specimens for research. The participants will be enrolled prior to the surgery, or they may be enrolled retrospectively and asked to share pathology specimens and slides previously collected that are no longer required for their medical care. Participants will be recruited from surgical protocols at the National Institutes of Health (NIH) Clinical Center or from other participating sites.
  * Part 2: Participants who have agreed to share surgical waste material may be asked to provide additional blood, saliva, and/or oral swabs. In addition, oral mucosal or skin biopsies may be obtained from adult participants aged 18 and older.
* No investigational or experimental therapy will be given as part of this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 3 and older.
* Able to provide their own consent, or for minors, a parent or guardian is able to consent on their behalf.
* Diagnosis of a condition of the head and neck for which removal of biological specimens was indicated for clinical care or for research purposes under a separate Review Board (IRB) approved protocol.
* Ability of subject (or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Part 1:

  --Are unwilling to share waste specimens for research purposes
* Part 2: Additional exclusion criteria for the Part 2 prospective sample collection part of this protocol these criteria may be assessed prior to collection of the samples but will not affect overall eligibility for the trial (i.e., Part 1):

  * have active symptomatic major organ disorders that would increase the risk of biopsy for research, including but not limited to bleeding disorders, ischemic heart disease, a recent myocardial infarction, active congestive heart failure or severe pulmonary dysfunction
  * have specific medical condition, such as a bleeding tendency where additional biopsies or phlebotomy procedures may increase the participants risk in participating. This will be determined at the discretion of the principal investigator
  * Individuals under the age of 18 are excluded from oral mucosal biopsies and skin biopsies

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants in this protocol will be a population with serious head and neck disorders, including cancer, and are anticipated to have a large number of adverse events completely unrelated to this protocol. Adverse events that are unrelated to the research under this protocol will not be reported to the IRB immediately or at the time of CR.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
To created a biorepository of diseased and normal tissue specimens for research purposes | 06/03/2026
  The primary endpoint of this study is the creation of a head and neck biorepository from both surgical waste material and prospectively collected blood, saliva, oral swabs, oral mucosa biopsy and skin biopsy specimens.

SECONDARY OUTCOMES:
To share repository specimens with other approved NIH protocols to conduct analysis of cellular, molecular, genetic and genomic biology of normal processes and disorders of the ENT. | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Clint T Allen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital Broadway Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital Bayview, Baltimore, Maryland
  - Johns Hopkins Hospital Greenspring, Baltimore, Maryland
  - Johns Hopkins Suburban Hospital, Bethesda, Maryland
  - Johns Hopkins Otolaryngology Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cancer Genome Atlas Network. Comprehensive genomic characterization of head and neck squamous cell carcinomas. Nature. 2015 Jan 29;517(7536):576-82. doi: 10.1038/nature14129. PMID 25631445
- [Background] Monasta L, Ronfani L, Marchetti F, Montico M, Vecchi Brumatti L, Bavcar A, Grasso D, Barbiero C, Tamburlini G. Burden of disease caused by otitis media: systematic review and global estimates. PLoS One. 2012;7(4):e36226. doi: 10.1371/journal.pone.0036226. Epub 2012 Apr 30. PMID 22558393
- [Background] Smith KA, Orlandi RR, Rudmik L. Cost of adult chronic rhinosinusitis: A systematic review. Laryngoscope. 2015 Jul;125(7):1547-56. doi: 10.1002/lary.25180. Epub 2015 Jan 30. PMID 25640115
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-DC-0051.html